CLINICAL TRIAL: NCT01321671
Title: The Pharmacokinetics Of Pregabalin Controlled Release Formulation In Fed State Compared To The Controlled Release And Immediate Release Formulations In The Fasted State
Brief Title: Investigation Of Absorption And Pharmacokinetics Of A Single Dose Of Controlled Release Pregabalin Tablet Administered Fasted In The Evening or Immediately Following A 600-750 Calorie Evening Meal As Compared To Single Dose Of Immediate Release Pregabalin Capsule In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0081228
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2011-06

CONDITIONS: Healthy
Keywords: pregabalin; pharmacokinetics; bioavailability; bioequivalence
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pregabalin controlled release, 330 mg, 600- 750 calorie (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg, 600- 750 calorie
- Pregabalin controlled release, 330 mg, fasted (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg, fasted
- Pregabalin immediate release, 300 mg (Other)
  Interventions: Drug: Pregabalin immediate release, 300 mg

INTERVENTIONS:
Drug: Pregabalin controlled release, 330 mg, 600- 750 calorie — A single oral dose of 330 mg controlled release tablet administered following a 600 to 750 calorie evening meal
  Arms: Pregabalin controlled release, 330 mg, 600- 750 calorie
Drug: Pregabalin controlled release, 330 mg, fasted — A single oral dose of 330 mg controlled release tablet administered fasted in the evening
  Arms: Pregabalin controlled release, 330 mg, fasted
Drug: Pregabalin immediate release, 300 mg — A single oral dose of 300 mg immediate release capsule administered in the evening
  Arms: Pregabalin immediate release, 300 mg

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of a single dose of a pregabalin controlled release (CR) tablet administered fasted in the evening relative to a single dose of the CR tablet administered immediately following a 600 to 750 calorie evening meal. The single dose pharmacokinetics of the pregabalin CR administered fed or fasted will also be compared to the single dose pharmacokinetics of the pregabalin immediate release (IR) capsule. In addition, the safety and tolerability of these 3 treatments will be evaluated.

DETAILED DESCRIPTION:
Evaluate the absorption, pharmacokinetics, safety/tolerability of a single dose of a pregabalin CR tablet under various conditions as compared to single dose of pregabalin IR capsule

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Illicit drug use
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve from 0 to infinity (AUCinf) and peak concentrations (Cmax) for assessment of equivalence between controlled released (CR) fed and CR fasted | 3 days
Area under the curve from 0 to infinity (AUCinf) for assessment of equivalence between the controlled release treatments and the immediate release treatment | 3 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Chew ML, Plotka A, Alvey CW, Pitman VW, Alebic-Kolbah T, Scavone JM, Bockbrader HN. Pharmacokinetics of pregabalin controlled-release in healthy volunteers: effect of food in five single-dose, randomized, clinical pharmacology studies. Clin Drug Investig. 2014 Sep;34(9):617-26. doi: 10.1007/s40261-014-0211-4. PMID 25078976
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081228&StudyName=Investigation%20Of%20Absorption%20And%20Pharmacokinetics%20Of%20A%20Single%20Dose%20Of%20Controlled%20Release%20Pregabalin%20Tablet%20Administered%20Fasted%20In%20The%20Eveni